CLINICAL TRIAL: NCT01828463
Title: An International, Multicentre, Randomised, Open-label, No-treatment Controlled, Parallel-group, Dose-response Study to Investigate the Effect of Once Daily Nitisinone on 24-hour Urinary Homogentisic Acid Excretion in Patients With Alkaptonuria After 4 Weeks Treatment.
Brief Title: Dose Response Study of Nitisinone in Alkaptonuria
Acronym: SONIA1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Professor Lakshminarayan Ranganath, Consultant in Metabolic medicine, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UoL000928
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Alkaptonuria
MeSH Terms: conditions — Alkaptonuria | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- no treatment (No Intervention): comparrator
- Nitisinone 1mg (Experimental): interventional
  Interventions: Drug: Nitisinone
- Nitisinone 2mg (Experimental): interventional
  Interventions: Drug: Nitisinone
- Nitisinone 4mg (Experimental): interventional
  Interventions: Drug: Nitisinone
- Nitisinone 8mg (Experimental): interventional
  Interventions: Drug: Nitisinone

INTERVENTIONS:
Drug: Nitisinone — doses 1, 2, 4 & 8 mg plus no treatment arm
  Arms: Nitisinone 1mg; Nitisinone 2mg; Nitisinone 4mg; Nitisinone 8mg

SUMMARY:
SONIA 1 is an international, multicentre, randomised, open-label, no-treatment controlled, parallel group, dose-response study to investigate the effect of once daily nitisinone on 24-hour urinary homogentisic acid excretion in patients with alkaptonuria after 4-weeks treatment. They study will identify the optimal dose to decrease urine homogentisic acid to near normal levels.

ELIGIBILITY:
Inclusion criteria

A subject must fulfil the following criteria in order to be included in the study:

1. Diagnosis of alkaptonuria verified by documented elevated urinary homogentisic acid excretion.
2. Age ≥18 years.
3. Willing and able to visit the investigational site for study visits.
4. Signed written informed consent obtained.

Exclusion criteria

The presence of any of the following will exclude a subject from inclusion in the study:

1. Non-alkaptonuria causes of ochronosis.
2. Currently pregnant or lactating.
3. Known allergy to nitisinone or any of the constituents of the investigational product.
4. Use of a protein-restricted diet
5. Dietary habits or use of homeopathic therapies that interfere with tyrosine catabolism.
6. Current keratopathy, contact lens use or uncontrolled glaucoma.
7. Current malignancy.
8. Uncontrolled hypertension (blood pressure greater than 180 systolic or greater than 95 diastolic).
9. Electrocardiogram changes indicative of myocardial infarction, arrhythmia, tachycardia, bradycardia, left bundle branch block.
10. Chest radiographic abnormalities, including an infiltrative, mass, congestive heart failure, embolism, atelectasis.
11. Serum potassium < 3.0 mmol/L.
12. eGFR < 60 mL/min.
13. Any hepatic enzymes greater than 3 x upper limit of normal.
14. Haemoglobin < 10.0 g/dL.
15. Platelets less than 100 x 109/L.
16. WBC less than 3.0 x 109/L.
17. ESR greater than 100 mm/h.
18. History of alcohol or drug abuse.
19. Participation in another clinical trial within 3 months of randomisation.
20. Treatment with nitisinone within 3 months of randomisation
21. Psychiatric illness or neurological disease that interferes with compliance or communication with health care personnel.
22. Any other medical condition which in the opinion of the investigator makes the subject unsuitable for inclusion.
23. Foreseeable inability to cooperate with given instructions or study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
dose of nitisinone that decreases urinary homogentisic acid to near normal | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: L Ranganath, Principal Investigator — Royal Liverpool & Broadgreen University Hospitals NHS Truts
Locations (1):
- Royal Liverpool Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] Milan AM, Hughes AT, Davison AS, Khedr M, Rovensky J, Psarelli EE, Cox TF, Rhodes NP, Gallagher JA, Ranganath LR. Quantification of the flux of tyrosine pathway metabolites during nitisinone treatment of Alkaptonuria. Sci Rep. 2019 Jul 11;9(1):10024. doi: 10.1038/s41598-019-46033-x. PMID 31296884
- [Derived] Ranganath LR, Milan AM, Hughes AT, Dutton JJ, Fitzgerald R, Briggs MC, Bygott H, Psarelli EE, Cox TF, Gallagher JA, Jarvis JC, van Kan C, Hall AK, Laan D, Olsson B, Szamosi J, Rudebeck M, Kullenberg T, Cronlund A, Svensson L, Junestrand C, Ayoob H, Timmis OG, Sireau N, Le Quan Sang KH, Genovese F, Braconi D, Santucci A, Nemethova M, Zatkova A, McCaffrey J, Christensen P, Ross G, Imrich R, Rovensky J. Suitability Of Nitisinone In Alkaptonuria 1 (SONIA 1): an international, multicentre, randomised, open-label, no-treatment controlled, parallel-group, dose-response study to investigate the effect of once daily nitisinone on 24-h urinary homogentisic acid excretion in patients with alkaptonuria after 4 weeks of treatment. Ann Rheum Dis. 2016 Feb;75(2):362-7. doi: 10.1136/annrheumdis-2014-206033. Epub 2014 Dec 4. PMID 25475116